CLINICAL TRIAL: NCT05485233
Title: Evaluation of Redscar © Application for Detection and Monitoring Potentially Infected Surgical Wounds: a Quasy-experimental Study Protocol
Brief Title: Redscar © Application for Detection of Infected Surgical Wounds
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hospital Son Espases (Other)
Collaborators: University of the Balearic Islands (Other); Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Responsible Party: Principal Investigator, Juan José Segura, Principal Investigator, Hospital Son Espases
Other Study IDs: IB4100/20 PI
Record Dates: First submitted 2022-07-01; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Surgical Wound Infection; Surgical Wound; Surgical Site Infection
Keywords: Surgical wound infection; Telematic follow-up; i-health
MeSH Terms: conditions — Surgical Wound Infection; Surgical Wound

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Presencial: At day 3th and 10th after surgery, each patient will undergo face-to-face examination of their surgical wound by a physician or a nurse, who will confirme the presence or absence of complications and they will fill in the questionnarie to compare the reponses with the aplication
- Telematic: At day 3th and 10th after surgery, each patient will upload an image of the surgical wound via RedScar© aplication using their own smartphone device. RedScar© aplication will evaluate the risk of complications of the surgical wound and will assign patients to 2 different groups: potential complications requiring new consultation or satisfactory evolution and discharge.
  Interventions: Device: REDSCAR App

INTERVENTIONS:
Device: REDSCAR App — Patients will be discharged after surgery at the time it is considered by the responsible physician. Prior to discharge, patients taking part in the study will follow the same protocol as any other patient treated in our institution. Written consent will be signed after complete explanation of the study protocol by the researcher at this moment. The patient will download the RedScar© application and the researcher will explain how it works and how to answer all the questions about the wound (redness, pain).
  At day 3th and 10th after surgery, each patient will upload an image of the surgical wound via RedScar© aplication using their own smartphone device. RedScar© aplication will evaluate the risk of complications of the surgical wound and will assign patients to 2 different groups: potential complications requiring new consultation or satisfactory evolution and discharge.
  Groups: Telematic

SUMMARY:
Surgical site infection (SSI) is the second cause of healthcare-associated infections (HAIs). Its appearance increase mobidity and post-operatice hospital stays, increasing costs aswell, although its one of the most preventable HAI.

The diagnosis and detection of SSI is usually carried out late by non-especialists once the patient has consulted to the emergency services or primary care with an already obvious infections. This raise both the direct and indirect costs and saturaties the emergency department and primary care, while delays treatment and increase disconfort and morbidity.

A smart phone aplication (RedScar© ) was developped in order to detect and monitor wound infection remotely based on an automated algorithm with no medical intervention.This app allows the patient to upload a photography and answer a short questionary, the aplication will then give a diagnosis of possible infection and recommendations.

This study is the first one to use a smartphone-based automatic aplication on real patients to diagnosis wound infection . This is a prospective, single-institution not randomized quasy-experimental study protocol. The study design and protocol were reviewed and approved by Research Ethics Committee of the Balearic Islands (CEI-IB).

This paper is part of the R+D+i Project PID2020-113870GB-I00- "Desarrollo de herramientas de Soft Computing para la Ayuda al Diagnóstico Clínico y a la Gestión de Emergencias (HESOCODICE)", funded by MCIN/AEI/10.13039/501100011033/.

ELIGIBILITY:
Inclusion Criteria:

* Signature of written consent.
* Age over 18 years.
* Emergency and scheduled surgery inpatients who have undergone abdominal surgery using staples to close the wound.
* Access to an android-based smartphone device, able to download the app and understand its management.
* Possibility of in person revision on the tenth postoperative day. Exclusion criteria
* Patients who do not have access to a compatible Smartphone or who are not able to use the app correctly (not being familiar with mobile devices or inability to understand how the app works or the questions asked).
* No written consent.
* Impossibility of personal revision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 30 emergency and scheduled surgery inpatients who are adults (over age 18 or with an authorization from mother/father/guardian) and have undergone abdominal laparotomy closed with staples will be screened for eligibility. Potentially eligible patients will be selected and documented as included, missed, rejected or excluded. Written consent will be obtained by the research team.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of RedScar© application to detect surgical infection compared to the face-to-face review. | 1 month
  Receiver operating characteristic (ROC) curve analysis will be used to identify the optimal cut-off value of Red Proportion in surgical infection screening with maximum sensitivity and specificity.
Number of participants with related adverse events as assessed by CTCAE v4.0 | 1 month

SECONDARY OUTCOMES:
Evaluate the satisfaction of the patients with the telematic care with the RedScar© app. | 1 month
  e satisfaction of the patients with the telematic care with the RedScar© app through the Telemedicine Satisfaction Questionnaire developed and validated by Yip MP et al. and on similar studies

CONTACTS AND LOCATIONS:
Overall Officials: Juan José Segura-Sampedro, Principal Investigator — Son Espases University Hospital
Locations (1):
- University Hospital Son Espases, Palma de Mallorca, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Global Guidelines for the Prevention of Surgical Site Infection. Geneva: World Health Organization; 2018. Available from http://www.ncbi.nlm.nih.gov/books/NBK536404/ PMID 30689333
- [Result] González-Hidalgo M, Moyà-Alcover G, Munar M, Bibiloni P, Craus-Miguel A, González-Argenté X, et al. Detection and Automatic Deletion of Staples in Images of Wound of Abdominal Surgery for m-Health Applications. In: Lecture Notes in Computational Vision and Biomechanics. 2019. p. 219-29. Available from: http://link.springer.com/10.1007/978-3-030-32040-9_23
- [Result] Healthcare-associated infections: surgical site infections - Annual Epidemiological Report for 2017 [Internet]. [cited 2022 Feb 27]. Available from: https://www.ecdc.europa.eu/en/publications-data/healthcare-associated-infections-surgical-site-infections-annual-1
- [Result] Yip MP, Chang AM, Chan J, MacKenzie AE. Development of the Telemedicine Satisfaction Questionnaire to evaluate patient satisfaction with telemedicine: a preliminary study. J Telemed Telecare. 2003;9(1):46-50. doi: 10.1258/135763303321159693. PMID 12641893
- [Result] Segura-Sampedro JJ, Rivero-Belenchon I, Pino-Diaz V, Rodriguez Sanchez MC, Pareja-Ciuro F, Padillo-Ruiz J, Jimenez-Rodriguez RM. Feasibility and safety of surgical wound remote follow-up by smart phone in appendectomy: A pilot study. Ann Med Surg (Lond). 2017 Jul 18;21:58-62. doi: 10.1016/j.amsu.2017.07.040. eCollection 2017 Sep. PMID 28794868
- [Derived] Craus-Miguel A, Munar M, Moya-Alcover G, Contreras-Nogales AM, Gonzalez-Hidalgo M, Segura-Sampedro JJ. Enhancing Surgical Wound Monitoring: A Paired Cohort Study Evaluating a New AI-Based Application for Automatic Detection of Potential Infections. J Clin Med. 2024 Dec 23;13(24):7863. doi: 10.3390/jcm13247863. PMID 39768786
- See also: Healthcare-associated infections: surgical site infections - Annual Epidemiological Report for 2017 — https://www.ecdc.europa.eu/en/publications-data/healthcare-associated-infections-surgical-site-infections-annual-1